CLINICAL TRIAL: NCT03324750
Title: Long-term Corticosteroid Use and Lifestyle Advices: A Qualitative Analysis of the Difficulties Encountered by Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0330
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-10

CONDITIONS: Patients Traited by Long Term Corticotherapy
Keywords: corticotherapy; qualitative study; therapeutic education; lifestyle change; diet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Nearly 1% of the population is currently treated with long-term corticosteroid therapy. When corticosteroids are introduced, patient information concerning the adverse effects and the modalities of prevention by the lifestyle changes is usually proposed. However, studies have shown an imperfect acquisition of this information about treatment and prevention of adverse effects, as well as a difficult implementation on diet and physical activity advices. In this study, the investigators aimed to evaluate the difficulties encountered by patients with dietary advice in the context of long-term corticosteroids use in order to optimize care, drug adherence and the quality of life of patients.

Methods: the investigators will recruite adult patients from general medicine and rheumatology practice and treated by long-term corticosteroids (≥ 3 months, ≥ 5mg/day). the investigators will perform a qualitative analysis in a semi-directed interview.

DETAILED DESCRIPTION:
Prospective Qualitative Study Carried out among patients followed in rheumatology and in general medical practice.

For each voluntary patient, a semi-directed interview was carried out in a consultation room after obtaining his agreement.

The same investigator used a single guide and conducted all the interviews based on open-ended questions.

At the end of the interviews, the entire recorded audio data was converted in written form before being analysed thematically.

Data were analysed using a Fisher's exact test for categorical variables (presented as frequencies and percentages), and using a non-parametric Mann-Whitney test for continuous variables (presented as the median and interquartile range, IQR).

ELIGIBILITY:
Inclusion Criteria:

* adult patients taking corticosteroids at an average dose ≥ 5 mg/day of equivalent prednisone over a period ≥ 3 months.

Exclusion Criteria:

* major memory impairment or language barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by long-term corticotherapy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
the difficulties encountered by patient in relation to the health and dietary advice given by physicians in the context of long term corticodteroid use | 1 day
  To determine the difficulties encountered by patient in relation to the health and dietary advice given by physicians in the context of long term corticodteroid use

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Lapeyronie, Montpellier, France